CLINICAL TRIAL: NCT03792516
Title: A Phase I Proof-of-Concept Study of Artesunate Ointment for the Treatment of Patients With High-Grade Vulvar Intraepithelial Neoplasia (HSIL VIN 2/3)
Brief Title: Artesunate Ointment for the Treatment of High Grade Vulvar Intraepithelial Neoplasia (HSIL VIN2/3)
Acronym: ART-VIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Frantz Viral Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J18169; IRB00196703 (Other: Johns Hopkins Medicine); IRB 19 1353 (Other: Cleveland Clinic Foundation)
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Vulvar Dysplasia; HPV-Related Vulvar Intraepithelial Neoplasia; Preinvasive Vulvar Disease; Vulva Intraepithelial Neoplasia; Vulvar Diseases
Keywords: artesunate; pre-invasive disease; treatment; alternative; non-surgical; cancer prevention
MeSH Terms: conditions — Vulvar Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Artesunate ointment 40%, 1 cycle (Experimental): Patients enrolled in this treatment group will receive one 5-day cycle of artesunate ointment applied topically to the vulva at week 0.
  Interventions: Drug: artesunate ointment 40%
- Artesunate ointment 40%, 2 cycles (Experimental): Patients enrolled in this treatment group will receive two 5-day cycles of artesunate ointment applied topically to the vulva at weeks 0 and 2.
  Interventions: Drug: artesunate ointment 40%
- Artesunate ointment 40%, 3 cycles (Experimental): Patients enrolled in this treatment group will receive three 5-day cycles of artesunate ointment applied topically to the vulva at weeks 0, 2, and 4.
  Interventions: Drug: artesunate ointment 40%

INTERVENTIONS:
Drug: artesunate ointment 40% — artesunate formulated as an ointment to be applied topically to the vulva

SUMMARY:
This is a Phase I, proof-of-concept treatment study to evaluate the safety, tolerability and feasibility of topical artesunate ointment to treat high grade vulvar intraepithelial neoplasia (HSIL VIN2/3).

DETAILED DESCRIPTION:
Phase I open-label dose escalation study of topical artesunate, formulated as ointment, in the treatment of adult females with biopsy-confirmed HSIL VIN2/3. Fifteen (15) subjects will undergo up to a total of three cycles of topical artesunate. The first cycle will be initiated on Day 0, the second at Week 2, and the third and final cycle at week 4.

Primary Objective:

To evaluate the safety and tolerability of artesunate ointment applied topically on VIN2/3 lesions

To measure the effect of artesunate ointment on histologic regression of HSIL/VIN2/3 to VIN1 or less, confirmed by a colposcopically-directed biopsy, at study week 15.

ELIGIBILITY:
Inclusion Criteria:

* Colposcopically-directed biopsy diagnosis of high-grade vulvar dysplasia (VIN2, VIN3, VIN2/3, HSIL), including both new and recurrent disease.
* Females of childbearing potential: negative urine pregnancy test
* Ability to provide informed consent
* Ability to collaborate with planned follow-up (transportation, compliance history, etc.)
* Use of contraception through the study exit visit (week 28)

Exclusion Criteria:

* Concomitant use of any topical immune modulating agents e.g. imiquimod, Aldara ®
* Cluster of differentiation 4 (CD4) count < 200 at the time of screening for eligibility.
* Unable to provide informed consent
* Currently receiving systemic chemotherapy or radiation therapy for another cancer.
* Pregnant females
* Concurrent dermatological disorders involving the vulva (i.e., herpes, ulceration secondary to Crohn's disease) or vulvar dermatosis (i.e., lichen planus, lichen sclerosus, or lichen simplex chronicus);
* Women weighing less than 50 kg

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for vulvar intraepithelial neoplasia, therefore it is only offerred to women.
Enrollment: 15 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of artesunate ointment applied topically on VIN2/3 lesions as assessed by number of participants experiencing serious adverse events or dose-limiting toxicities | 15 weeks
  Number of participants with study-related serious adverse events or dose-limiting toxicities assessed using Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) criteria

SECONDARY OUTCOMES:
Effect of artesunate ointment as assessed by number of participants with regression to VIN1 or less at week 15 | 15 weeks
  Number of participants with histologic regression of HSIL/VIN2/3 to VIN1 or less on colposcopically-directed biopsy, at study week 15 after receiving artesunate ointment therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Trimble, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation - Main Campus, Cleveland, Ohio
  - Cleveland Clinic - Hillcrest Hospital, Mayfield Heights, Ohio

IPD SHARING:
Plan to Share IPD: No